CLINICAL TRIAL: NCT03436199
Title: A 3-arm, Multicenter, Double-blind, Placebo-controlled, Randomized Study to Assess the Efficacy and Safety of ADS-5102 Amantadine Extended Release Capsules in Multiple Sclerosis Patients With Walking Impairment
Brief Title: Safety and Efficacy of ADS-5102 in Multiple Sclerosis Patients With Walking Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adamas Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADS-AMT-MS301
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Results first posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Walking Impairment; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ADS-5102, 137 mg (Experimental): ADS-5102, administered once daily at bedtime from Week 4 through Week 16
  Interventions: Drug: ADS-5102, 137 mg
- ADS-5102, 274 mg (Experimental): ADS-5102, administered once daily at bedtime from Week 4 through Week 16
  Interventions: Drug: ADS-5102, 274 mg
- Placebo (Other): placebo, administered once daily at bedtime from Week 4 through Week 16
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ADS-5102, 137 mg — Oral capsules
  Other Names: ADS-5102; amantadine extended release
  Arms: ADS-5102, 137 mg
Drug: ADS-5102, 274 mg — Oral capsules
  Other Names: ADS-5102; amantadine extended release
  Arms: ADS-5102, 274 mg
Other: Placebo — Oral capsules
  Arms: Placebo

SUMMARY:
This study assessed the efficacy and safety of ADS-5102 (at daily doses of 137 mg or 274 mg) compared with placebo in MS patients with walking impairment.

DETAILED DESCRIPTION:
This was a multicenter, 3-arm, randomized, placebo-controlled, double-blind, parallel-group study of ADS-5102 (amantadine) extended release capsules in MS subjects with walking impairment. The study consisted of a screening period (up to 3 weeks), a single-blind placebo run-in period (4 weeks; during which subjects were blinded to treatment), and a double-blind treatment period (12 weeks).

For at least 30 days prior to screening, all subjects were to have received a stable regimen of MS medications, both disease-modifying and symptomatic; these medications were to continue at the same doses and regimens for the duration of the subjects' participation in the study, to the extent compatible with good neurological care. Subjects were not to have used amantadine, dalfampridine, or any 4 aminopyridine or 2,4 diaminopyridine preparation within 30 days prior to screening.

Consented subjects who completed the screening period were to undergo a 4-week single-blind placebo run-in period during which they received placebo as 2 capsules once daily at bedtime.

Subjects who completed the single-blind placebo run-in period and continued to meet study eligibility criteria were randomized with equal probability to 1 of 3 treatment groups: placebo or ADS-5102 at a final dose of 137 mg/day or 274 mg/day. Study drugs were administered as 2 capsules once daily at bedtime.

Subjects were to return to the clinic for safety and efficacy assessments at Week 0 and Week 2 prior to randomization and at Weeks 4 (randomization and baseline visit), 6 (only safety), 8, 12, and 16 after randomization. In addition, telephone visits for safety assessments were conducted at Weeks 5 and 7. Subjects who withdrew from the study before Week 16 were to have an early termination visit that included safety follow-up and efficacy assessments, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Signed a current IRB-approved informed consent form
* Male or female subjects between 18 and 70 years of age, inclusive, at the time of Screening
* Confirmed diagnosis of MS according to the 2017 McDonald criteria
* Current medication regimen must be stable for at least 30 days prior to screening, and subject must be willing to continue the same dosing regimen for the duration of study participation
* Maximum Expanded Disability Status Scale (EDSS) score during screening of 6.5
* Stable physical activity level (inclusive of prescribed physical therapy) for at least 30 days prior to screening and willing to continue without change for the duration of study participation
* A score on each of two completed screening T25FW tests between 8 and 45 seconds, inclusive

Exclusion Criteria:

* Documented inability to tolerate amantadine
* Clinically significant MS relapse with onset less than 30 days prior to screening
* Receipt of dalfampridine (or any 4-aminopyridine or 2,4-diaminopyridine preparation) or amantadine within 30 days prior to screening
* History of seizures within 3 years prior to screening
* History of hallucinations (visual, auditory, or any other type) within 3 years prior to screening
* History of bipolar disorder, schizophrenia, or psychosis, regardless of treatment
* For subjects with a history of major depressive disorder, the presence of active depressive symptoms that, in the opinion of the investigator, would affect the subject's ability to complete study assessments, or which would not be in the subject's best interest to participate in the study
* Presence of orthostatic hypotension at screening: a decrease in systolic blood pressure (at least 20 mm Hg) or diastolic blood pressure (at least 10 mm Hg) within 3 minutes of the subject standing up, compared to pressures obtained while sitting
* If female, is pregnant or lactating
* If a sexually active female, is not surgically sterile or at least 2 years post-menopausal, or does not agree to utilize a highly effective hormonal method of contraception (an IUD, or vasectomized male partner is also acceptable), in combination with a barrier method, from screening through at least 4 weeks after the completion of study treatment. If a sexually active male, does not agree to utilize condoms from screening through at least 4 weeks after the completion of study treatment.
* Treatment with an investigational drug or device within 30 days prior to screening
* Treatment with an investigational biologic within 6 months or 5 half-lives, whichever is longer, prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Director, Study Director — Adamas Pharmaceuticals
Locations (82):
- United States (76):
  - Adamas Clinical Site, Cullman, Alabama
  - Adamas Clinical Site, Phoenix, Arizona
  - Adamas Clinical Site, Scottsdale, Arizona
  - Adamas Clinical Site, Tucson, Arizona
  - Adamas Clinical Site, Carlsbad, California
  - Adamas Clinical Site, Fresno, California
  - Adamas Clinical Site, Fullerton, California
  - Adamas Clinical Site, Long Beach, California
  - Adamas Clinical Site, Newport Beach, California
  - Adamas Clinical Site, Sacramento, California
  - Adamas Clinical Site, Aurora, Colorado
  - Adamas Clinical Site, Colorado Springs, Colorado
  - Adamas Clinical Site, Denver, Colorado
  - Adamas Clinical Site, Fort Collins, Colorado
  - Adamas Clinical Site, Fairfield, Connecticut
  - Adamas Clinical Site, New London, Connecticut
  - Adamas Clinical Site, Washington D.C., District of Columbia
  - Adamas Clinical Site, Maitland, Florida
  - Adamas Clinical Site, Miami, Florida
  - Adamas Clinical Site, Naples, Florida
  - Adamas Clinical Site, Orlando, Florida
  - Adamas Clinical Site, Ormond Beach, Florida
  - Adamas Clinical Site, Palm Coast, Florida
  - Adamas Clinical Site, Port Charlotte, Florida
  - Adamas Clinical Site, Sarasota, Florida
  - Adamas Clinical Site, Tampa, Florida
  - Adamas Clinical Site, Vero Beach, Florida
  - Adamas Clinical Site, Atlanta, Georgia
  - Adamas Clinical Site, Savannah, Georgia
  - Adamas Clinical Site, Northbrook, Illinois
  - Adamas Clinical Site, Indianapolis, Indiana
  - Adamas Clinical Site, Kansas City, Kansas
  - Adamas Clinical Site, Lenexa, Kansas
  - Adamas Clinical Site, Overland Park, Kansas
  - Adamas Clinical Site, Foxborough, Massachusetts
  - Adamas Clinical Site, Lexington, Massachusetts
  - Admas Clinical Site, Detroit, Michigan
  - Adamas Clinical Site, Farmington Hills, Michigan
  - Adamas Clinical Site, Golden Valley, Minnesota
  - Adamas Clinical Site, Kansas City, Missouri
  - Adamas Clinical Site, St Louis, Missouri
  - Adamas Clinical Site, Great Falls, Montana
  - Adamas Clinical Site, Lincoln, Nebraska
  - Adamas Clinical Site, Omaha, Nebraska
  - Adamas Clinical Site, Las Vegas, Nevada
  - Adamas Clinical Site, Albuquerque, New Mexico
  - Adamas Clinical Site, Amherst, New York
  - Adamas Clinical Site, Lake Success, New York
  - Adamas Clinical Site, New York, New York
  - Adamas Clinical Site, Patchogue, New York
  - Adamas Clinical Site, Plainview, New York
  - Adamas Clinical Site, Rochester, New York
  - Adamas Clinical Site, Staten Island, New York
  - Adamas Clinical Site, Charlotte, North Carolina
  - Adamas Clinical Site, Raleigh, North Carolina
  - Adamas Clinical Site, Centerville, Ohio
  - Adamas Clinical Site, Cleveland, Ohio
  - Adamas Clinical Site, Columbus, Ohio
  - Adamas Clinical Site, Oklahoma City, Oklahoma
  - Adamas Clinical Site, Portland, Oregon
  - Adamas Clinical Site, Philadelphia, Pennsylvania
  - Adamas Clinical Site, Charleston, South Carolina
  - Adamas Clinical Site, Greer, South Carolina
  - Adamas Clinical Site, Old Point Station, South Carolina
  - Adamas Clinical Site, Spartanburg, South Carolina
  - Adamas Clinical Site, Cordova, Tennessee
  - Adamas Clinical Site, Franklin, Tennessee
  - Adamas Clinical Site, Johnson City, Tennessee
  - Adamas Clinical Site, Houston, Texas
  - Adamas Clinical Site, Round Rock, Texas
  - Adamas Clinical Site, Salt Lake City, Utah
  - Adamas Clinical Site, Newport News, Virginia
  - Adamas Clinical Site, Norfolk, Virginia
  - Adamas Clinical Site, Kirkland, Washington
  - Adamas Clinical Site, Seattle, Washington
  - Adamas Clinical Site, Milwaukee, Wisconsin
- Canada (6):
  - Adamas Clinical Site, Edmonton, Alberta
  - Adamas Clinical Site, Lethbridge, Alberta
  - Adamas Clinical Site, Burnaby, British Columbia
  - Adamas Clinical Site, Greenfield Park, Quebec
  - Adamas Clinical Site, Montreal, Quebec
  - Adamas Clinical Site, Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- ADS-5102 137 mg: ADS-5102, 137 mg: Oral capsules to be administered once daily at bedtime
- ADS-5102 274 mg: ADS-5102, 274 mg: Oral capsules to be administered once daily at bedtime
- Placebo: placebo capsules
  Placebo: Oral capsules to be administered once daily at bedtime
Period: Overall Study
Arm/Group | ADS-5102 137 mg | ADS-5102 274 mg | Placebo
Started | 187 | 185 | 186
Completed | 165 | 132 | 174
Not Completed | 22 | 53 | 12
Not completed — Adverse Event | 15 | 40 | 7
Not completed — Withdrawal by Subject | 4 | 10 | 3
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Could not return to clinic | 1 | 0 | 0
Not completed — Withdrawn per physician | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADS-5102 137 mg | ADS-5102 274 mg | Placebo | Total
Number analyzed (Participants) | 187 | 185 | 186 | 558
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (9.13) | 54.0 (9.27) | 54.5 (9.75) | 54.4 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 124 | 128 | 377
  Male | 62 | 61 | 58 | 181
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 3
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 24 | 21 | 23 | 68
  White | 158 | 160 | 155 | 473
  More than one race | 1 | 0 | 3 | 4
  Unknown or Not Reported | 3 | 4 | 3 | 10
Time since diagnosis of multiple sclerosis [Mean (Standard Deviation); unit: years] | 15.99 (9.862) | 15.97 (9.655) | 15.85 (9.478) | 15.94 (9.649)

OUTCOME MEASURES:

1. Primary Outcome: Timed 25 Foot Walk (T25FW, Feet/Second): the Proportion of Subjects With a ≥ 20% Increase in Walking Speed (Measured by T25FW) From Baseline at Week 16 (Responder Analysis)
Description: The T25FW is a measure of lower extremity function. The subject is directed to a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The task is immediately administered again by having the subject walk back the same distance. For this outcome measure, the result is reported as speed (feet per second). Improvement is indicated by an increase in speed.
Time Frame: 16 weeks
Population: Intent-to-treat population
Measure: Number; unit: proportion of responders
Arm/Group | ADS-5102 137 mg | ADS-5102 274 mg | Placebo
Number analyzed (Participants) | 187 | 185 | 186
proportion of responders | 0.176 | 0.211 | 0.113
Statistical Analysis 1: Comparison: ADS-5102 137 mg vs Placebo; Test type: Superiority; p = 0.0811, Farrington-Manning score test; The Miettinen-Nurminen method was used to obtain the 95% confidence intervals; Risk Difference (RD) = 0.064, 95% CI 2-sided [-0.008 to 0.136]
Statistical Analysis 2: Comparison: ADS-5102 274 mg vs Placebo; Test type: Superiority; p = 0.0104, Farrington-Manning score test; The Miettinen-Nurminen method was used to obtain the 95% confidence intervals; Risk Difference (RD) = 0.098, 95% CI 2-sided [0.023 to 0.174]

2. Secondary Outcome: Timed 25 Foot Walk: Change From Baseline at Week 16
Description: The T25FW is a measure of lower extremity function. The subject is directed to a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The task is immediately administered again by having the subject walk back the same distance. For this outcome measure, the result is reported as or speed (feet per second). Improvement is indicated by an increase in speed.
Time Frame: 16 weeks
Population: Intent-to-treat: subjects with available data at Week 16
Measure: Least Squares Mean (Standard Error); unit: feet/second
Arm/Group | ADS-5102 137 mg | ADS-5102 274 mg | Placebo
Number analyzed (Participants) | 167 | 135 | 176
feet/second | 0.19 (0.034) | 0.19 (0.034) | 0.07 (0.033)
Statistical Analysis 1: Comparison: ADS-5102 137 mg vs Placebo; Test type: Superiority; p = 0.0162, Mixed Models Analysis; Mixed models analysis with repeated measures; Mean Difference (Net) = 0.12, 95% CI 2-sided [0.02 to 0.21], Standard Error of Mean 0.048
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority; p = 0.0142, Mixed Models Analysis; Mixed models analysis with repeated measures; Mean Difference (Net) = 0.12, 95% CI 2-sided [0.02 to 0.22], Standard Error of Mean 0.050

3. Secondary Outcome: Timed Up and Go (TUG): Change From Baseline at Week 16
Description: The TUG is a measure of lower extremity strength, balance, and coordination. The subject stands up from a chair, walks 3 meters then turns around and walks back to the chair to sit down. The result is reported in seconds. Improvement is indicated by negative change scores.
Time Frame: 16 weeks
Population: Intent-to-treat: subjects with available data at Week 16
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | ADS-5102 137 mg | ADS-5102 274 mg | Placebo
Number analyzed (Participants) | 168 | 136 | 176
seconds | -1.35 (0.384) | -0.60 (0.415) | -0.56 (0.377)
Statistical Analysis 1: Comparison: ADS-5102 137 mg vs Placebo; Test type: Superiority; p = 0.1424, Mixed Models Analysis; Mixed models analysis with repeated measures; Mean Difference (Net) = -0.79, 95% CI 2-sided [-1.85 to 0.27], Standard Error of Mean 0.538
Statistical Analysis 2: Comparison: ADS-5102 274 mg vs Placebo; Test type: Superiority; p = 0.9467, Mixed Models Analysis; Mixed models analysis with repeated measures; Mean Difference (Net) = -0.04, 95% CI 2-sided [-1.14 to 1.06], Standard Error of Mean 0.560

4. Secondary Outcome: 2-Minute Walk Test (2MWT): Change From Baseline at Week 16
Description: The 2MWT is a measure of lower extremity function. The subject is instructed to walk as far as possible in 2 minutes, and the distance is measured in meters. Improvement is indicated by positive change scores.
Time Frame: 16 weeks
Population: Intent-to-treat: subjects with available data at Week 16
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | ADS-5102 137 mg | ADS-5102 274 mg | Placebo
Number analyzed (Participants) | 167 | 136 | 176
meters | 6.306 (1.2422) | 5.692 (1.3537) | 2.163 (1.2158)
Statistical Analysis 1: Comparison: ADS-5102 137 mg vs Placebo; Test type: Superiority; p = 0.0176, Mixed Models Analysis; Mixed models analysis with repeated measures; Mean Difference (Net) = 4.143, 95% CI 2-sided [0.726 to 7.560], Standard Error of Mean 1.7389
Statistical Analysis 2: Comparison: ADS-5102 274 mg vs Placebo; Test type: Superiority; p = 0.0530, Mixed Models Analysis; Mixed models analysis with repeated measures; Mean Difference (Net) = 3.529, 95% CI 2-sided [-0.046 to 7.104], Standard Error of Mean 1.8196

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | ADS-5102 137 mg | ADS-5102 274 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/187 | 0/185 | 0/186
Serious Adverse Events (participants affected / at risk) | 5/187 | 11/185 | 1/186
Other Adverse Events (participants affected / at risk) | 105/187 | 140/185 | 90/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADS-5102 137 mg (N=187) | ADS-5102 274 mg (N=185) | Placebo (N=186)
Appendicitis (Infections and infestations) | 1 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 2 | 0
Facial spasm (Nervous system disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hallucinations, mixed (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADS-5102 137 mg (N=187) | ADS-5102 274 mg (N=185) | Placebo (N=186)
Oedema peripheral (General disorders) | 8 | 29 | 1
Dry mouth (Gastrointestinal disorders) | 6 | 25 | 2
Constipation (Gastrointestinal disorders) | 8 | 15 | 1
Urinary tract infection (Infections and infestations) | 7 | 16 | 19
Insomnia (Psychiatric disorders) | 3 | 13 | 0
Fall (Injury, poisoning and procedural complications) | 8 | 16 | 13
Nasopharyngitis (Infections and infestations) | 7 | 4 | 7
Dizziness (Nervous system disorders) | 5 | 8 | 4
Tremor (Nervous system disorders) | 2 | 8 | 1
Fatigue (General disorders) | 6 | 8 | 5
Peripheral swelling (General disorders) | 1 | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 7
Contusion (Injury, poisoning and procedural complications) | 3 | 7 | 4
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 7 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 6 | 2
Vision blurred (Eye disorders) | 2 | 8 | 1
Dry eye (Eye disorders) | 0 | 6 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 6 | 1
Sinusitis (Infections and infestations) | 1 | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 5 | 1
Headache (Nervous system disorders) | 4 | 5 | 4
Multiple sclerosis relapse (Nervous system disorders) | 2 | 5 | 3
Balance disorder (Nervous system disorders) | 1 | 5 | 0
Gait disturbance (General disorders) | 2 | 4 | 0
Hallucinations, visual (Psychiatric disorders) | 4 | 5 | 0
Anxiety (Psychiatric disorders) | 1 | 6 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5 | 3
Skin abrasion (Injury, poisoning and procedural complications) | 4 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Hypertension (Vascular disorders) | 2 | 5 | 3
Vertigo (Ear and labyrinth disorders) | 2 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT03436199/Prot_SAP_000.pdf